CLINICAL TRIAL: NCT00548431
Title: Phase II Study of Individual 6-mercaptopurine(6MP) Dose Increments in Children With Acute Lymphoblastic Leukemia (ALL) Receiving High-dose Methotrexate (HDM) and PEG-asparaginase
Brief Title: NOPHO ALL-2008 Pilot Study on Consolidation Therapy for Children and Adolescents With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO HDM-6MP pilot study
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Results first posted 2010-11-03 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Leukemia, Lymphocytic, Acute
Keywords: Leukemia, Lymphocytic, Acute [C04.557.337.428.511]; 6-mercaptopurine; methotrexate; asparaginase
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6 mercaptopurine arm (Experimental): All patients received basic daily 6MP (6-mercaptopurine) (25 mg/m^2) and in addition high-dose methotrexate(HDM) every 3rd week (3 times HDM in total) and PEG-asparaginase every 14th day. Patients increased the dose of 6MP 2 weeks after each HDM if if the myelotoxicity had been acceptable. This means 2 increments since the study stopped 2 weeks after the last HDM
  Interventions: Drug: 6-mercaptopurine

INTERVENTIONS:
Drug: 6-mercaptopurine — Standard dose 25 mg/m^2/day. Can be increased up to 75 mg/m^2/day if the myelosuppression is acceptable (ANC>0.5 T-count >50)
  Other Names: PURINETHOL

SUMMARY:
The present pharmacokinetic (PK)-pharmacodynamic (PD) study will explore the toxicity and antileukemic response during the initial 3 months of individualised therapy of children and young adults with acute lymphoblastic leukemia (ALL). The investigators will on an individual toxicity-titrated basis attempt to increase the dose intensity of the 6-mercaptopurine used in the two-months post-remission treatment phase of lower risk childhood ALL. This will be performed together with continuous PEG-ASP (every 2nd week) and interspersed HD-MTX (5 g/m^2) every 3rd week. Thus, the trial will also test the feasibility of this particular drug combination.

DETAILED DESCRIPTION:
In addition to the details above we will also explore

* the relationship of the post-HD-MTX MRD-levels with the dose of 6MP, TPMT-activity, DNA-6TGN, E-6TGN, E-MeMP, E-MTX, and presence of ASP-antibodies,
* the early development of anti-ASP antibodies during continuous PEG-ASP therapy.

The study could improve the understanding of the pharmacodynamics of the 6MP/HD-MTX interaction in combination with PEG-ASP.

ELIGIBILITY:
Inclusion Criteria:

* B-lineage ALL
* 1-17.9 years
* WBC <100, clinical remission obtained day 2
* Written consent to participation.

Exclusion Criteria:

* t(9;22)
* Hypodiploidy
* 11q23-aberrations
* TPMT-deficiency
* Intolerance to MTX or 6MP

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Study Chair — Pediatric Clinic II, RIgshospitalet, Copenhagen, DK-2100
Locations (3):
- Denmark (2):
  - Department of Pediatrics, Rigshospitalet, Copenhagen
  - Department of Pediatrics, University Hospital, Odense
- Department of Pediatrics, Drottning Sylvias Pediatric Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data published (Frandsen et al, Br J Haematol Oct 2011) Anonymised data on individual patients can be provided by study chair (kschmiegelow@rh.dk) including studyno, gender, age, thiopurine methyltransferase status, immunophenotype, white blood cell count at diagnosis, dose increments at time point 1 and 2 for dose adjustment, and dose-limiting toxicities

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients were recruited in 3 different countries. Recruitment period 12/01/2007 - 12/21/2008. All recruitments were done in departments of Pediatric Hematology/oncology
Groups:
- 6-mercaptopurine: All patients received basic 6-mercaptopurine and in addition high-dose methotrexate(HDM) at 3 week intervals ((3 3-week intervals) in total) and PEG-asparaginase at 2 week intervals(5 dosis in total) . Patients received dose increments of 6-mercaptopurine 14 days after High-dose methotrexate if the myelotoxicity was acceptable
Period: Overall Study
Arm/Group | 6-mercaptopurine
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 6-mercaptopurine
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (3)
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Region of Enrollment [Number; unit: participants]
  Denmark | 12
  Sweden | 21
  Finland | 5

OUTCOME MEASURES:

1. Primary Outcome: Toxicity of Treatment in Terms of Number of Participants With Serious Adverse Events or Adverse Events, Reported
Description: Number of participants following the protocol treatment for the full consolidation therapy with toxicity in this pilot study trying to individually titrate 6-mercaptopurine to the highest tolerable level during Consolidation.
Time Frame: 3 months ( 79 days )
Measure: Number; unit: Participants
Arm/Group | 6-mercaptopurine
Number analyzed (Participants) | 38
Participants | 26

2. Secondary Outcome: Incorporation of 6-thioguanine Nucleotides (6TGN) Into Leukocyte DNA, Development of Asparaginase Antibody Production
Description: Biweekly bloodsamples during the 3 months are analyzed for 6TGN incorporation into leucocyte DNA. In addition Methylated Mercaptopurine (MeMP) and Erythrocyte-Methotrexate level is measured
Time Frame: During the 3 months consolidation therapy
Reporting Status: Not Posted, anticipated posting 2018-02

ADVERSE EVENTS:
Time Frame: Adverse events were reported for each patient for a period of 3 months
Description: Adverse events were recorded in a bi-weekly questionaire to be filled by physician and patient/parents.
Arm/Group | 6-mercaptopurine
Serious Adverse Events (participants affected / at risk) | 26/38
Other Adverse Events (participants affected / at risk) | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-mercaptopurine (N=38)
Hypoglycemia (Hepatobiliary disorders) | 2 (2) — 2 patients had hypoglycemia due to liver toxicity. Not an unusual event during 6MP treatment, but somewhat early in the treatment. Both had to be hospitalized longer due to this adverse event.
neutropenic fever (Congenital, familial and genetic disorders) | 22 (30) — admission to hospital for neutropenic fever is expected during leukemia treatment in the consolidation phase. Usually patients are admitted for i.v. antibiotic treatment for 5-10 days depending on neutropenia and agent.
pancreatitis (Gastrointestinal disorders) | 1 (1) — grade 4 pancreatitis
PRES (Posterior Reversible Encephalopathy Syndrome) (Nervous system disorders) | 1 (1) — Hypertension and PRES in connection with High Dose Methotrexate.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6-mercaptopurine (N=38)
pain (Gastrointestinal disorders) | 23 (55) — pain is also expected during treatment of leukemia in childhool. Most common pain from abdomen or legs or mouth (stomatitis)
mucositis (Gastrointestinal disorders) | 22 (30) — Mucositis following chemotherapy-mostly high dose Methotrexate in combination with 6MP
nausea and vomiting (Gastrointestinal disorders) | 21 (68)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No